CLINICAL TRIAL: NCT04444232
Title: Cancer Communication Within Social Networks
Brief Title: Cancer Communication Within Hispanic Social Networks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: RG1001018; P30CA015704 (NIH); NCI-2020-04236 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 8182 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2020-06-19; First posted 2020-06-23 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health services research (educational video, survey) (Experimental): Participants view an educational video on cancer and cancer screening options over 12 minutes. Participants also complete a phone survey over 10-15 minutes before attending the video session and 2 months after the video session.
  Interventions: Other: Media Intervention; Other: Survey Administration

INTERVENTIONS:
Other: Media Intervention — View an educational video
Other: Survey Administration — Complete survey

SUMMARY:
This trial examines cancer communication within Hispanic social networks. Hispanics have the lowest colorectal cancer screening rate of any major ethnic group and health interventions are crucially needed among Hispanics. Patient decision aids are health communication interventions designed to provide patients with targeted health information and have shown to improve colorectal cancer screening rates among Hispanics. The goal of this study is to investigate, in a sample of Hispanics, how a colorectal cancer decision aid aimed at increasing individuals' colorectal cancer screening behavior has effects on their alters' intention to get screened for colorectal cancer.

DETAILED DESCRIPTION:
OUTLINE:

Participants view an educational video on cancer and cancer screening options over 12 minutes. Participants also complete a phone survey over 10-15 minutes before attending the video session and 2 months after the video session.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as "Hispanic" or "Latino"
* Have no family history of CRC
* Have no personal history of pre-cancerous (adenomatous) colonic polyps
* Have not had either an annual fecal occult blood test (FOBT) within the past year or colonoscopy within the last 10 years (defined as up-to-date with CRC screening by current United States [U.S.] Preventive Services Task Force recommendations)
* Have at least two family members, friends, or co-workers who are ages 50-75
* Alters will be eligible if they are ages 50-75

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2014-09-09 (Actual); Primary Completion 2015-02-10 (Actual); Study Completion 2015-03-09 (Actual)

PRIMARY OUTCOMES:
Patients' communication with their families, friends, and co-workers about colorectal cancer (CRC) screening | Up to 6 months
  Will be assessed using a single dichotomized question with two response options ('yes' or 'no'). CRC communication constitutes in-person conversation, email, phone, or post on social media (e.g., blog, Twitter, Facebook). Will also assess the characteristics of the alters by asking the patients two questions on social-tie dimensions: 1) contact frequency (never, rarely, sometimes, often, or very often) and 2) personal relationship (acquaintance , close friend , co-worker, relatives, or spouse).
Alters' intent to become screened for CRC in the next six months | Up to 6 months
  Intent will be assessed using a single categorical item with three response options (definitely planning to be screened, considering being screened, not considering being screened).

CONTACTS AND LOCATIONS:
Overall Officials: Linda Ko, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ko LK, Jang SH, Rodriguez E, Buta M, Ibarra G, Reuland D. Dissemination of colorectal cancer information among Hispanic patients and their social network. BMC Public Health. 2024 Sep 27;24(1):2616. doi: 10.1186/s12889-024-20095-7. PMID 39334118